CLINICAL TRIAL: NCT05755295
Title: Pilot Study Evaluating Feasibility and Acceptability of Horse Therapy for Children, Adolescents and Young Adults in Remission From Medulloblastoma and Describing the Evolution of Their Physical and Psychological Characteristics
Brief Title: Horse Therapy for Children, Adolescents and Young Adults in Remission From Medulloblastoma
Acronym: EQUI-HIPPO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/22/0218
Record Dates: First submitted 2023-02-22; First posted 2023-03-06 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Neuroblastoma
Keywords: hippotherapy; equitherapy
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- horse therapy (Experimental)
  Interventions: Other: horse therapy

INTERVENTIONS:
Other: horse therapy — equitherapy and hippotherapy once a week during 16 weeks

SUMMARY:
On average, each year in the former region, 60 new patients under the age of 18 are treated for a brain tumor, with an active post-treatment follow-up file of 350 patients. Because of the significant sequelae induced by the disease or the treatments, these patients will very often require rehabilitative care.

The interest of involving the horse in the population of patients cured of a medulloblastoma but with important physical and psychological after-effects is to be able to combine a therapy using animal mediation (equitherapy) and a rehabilitation therapy based on the three-dimensional movement of the horse (hippotherapy).

ELIGIBILITY:
Inclusion Criteria:

* complete remission of medulloblastoma and after 5 years of the end of treatment
* living within 30 km away the riding center and/or less than 1 hour of transport
* informed consent

Exclusion Criteria:

* Landsky score below 50% for minors until 16 years old and Karnofsky score below 50% for patients over 16 years
* major under juridical protection

Ages: 10 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
number of sessions performed | 16 weeks
  number of sessions equitherapy and hippotherapy performed

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Isabelle BERTOZZI, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No